CLINICAL TRIAL: NCT06835439
Title: Improving Access and Engagement in Spine Pain Rehabilitation - STEPPT Mixed Methods Pilot Study
Brief Title: Development of STEPPT
Acronym: STEPPT PILOT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Family Health Centers of San Diego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-24-0391; R01MD018937 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-19 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pain; Back Pain; Low Back Pain; Chronic Pain; Neck Pain
Keywords: Physical therapy; Rehabilitation; Hispanic; Health disparities; Health services; Healthcare utilization
MeSH Terms: conditions — Pain; Back Pain; Low Back Pain; Chronic Pain; Neck Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The primary purpose of this pilot study is to assess the feasibility, acceptability, and estimate effect size of the pilot STEPPT intervention for improving ethnic disparities in physical therapy referral and adherence between Hispanic and Non-Hispanic White patients with spine pain. The health services intervention design is a single site, mixed-methods pilot study using a non-randomized quasi-experimental pre-post design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPPT Intervention (Experimental): Participants in this arm will receive the pilot STEPPT intervention, which includes (1) education of providers and staff on disparities in referrals and the benefits of physical therapy for spine pain, (2) modifications to the EHR to automate physical therapy referral and delivery of culturally tailored patient education materials, and (3) enhanced patient health navigation to educate patients and address barriers to attending physical therapy for Hispanic patients with spine pain. The goal is to reduce ethnic disparities by improving physical therapy referral and adherence rates for Hispanic patients with spine pain.
  Interventions: Behavioral: STEPPT Pilot
- Standard Care (Control) (Active Comparator): Standard care during the 3-month baseline period, prior to implementing the STEPPT intervention, will be the active comparator arm. Ethnic disparities in referral and adherence rates will be compared between the 3-month baseline period and the 3-month intervention period to estimate the effect size of the pilot STEPPT intervention for reducing ethnic disparities in physical therapy referral and adherence outcomes.
  Interventions: Behavioral: Standard Care (Control)

INTERVENTIONS:
Behavioral: STEPPT Pilot — The pilot STEPPT intervention, which includes (1) education of providers and staff on disparities in referrals and the benefits of physical therapy for spine pain, (2) modifications to the EHR to automate physical therapy referral and delivery of culturally tailored patient education materials related to the physical therapy referral, and (3) enhanced patient health navigation to educate patients on physical therapy and address barriers to attending physical therapy for Hispanic patients with spine pain. Patient education materials were developed using evidence-based guidelines and were culturally and linguistically adapted for Hispanic patients with spine pain.
  Arms: STEPPT Intervention
Behavioral: Standard Care (Control) — Usual care (3-month baseline) includes no provider education, physician-initiated referrals and delivery of standard educational materials, and scheduling for physical therapy by the clinic referrals specialists using standard processes.
  Arms: Standard Care (Control)

SUMMARY:
This 6-month pilot study aims to assess the feasibility, acceptability, and estimate effect sizes of the pilot STEPPT intervention for addressing ethnic disparities in physical therapy referrals and adherence between Hispanic and Non-Hispanic White patients with spine pain. Feasibility and acceptability will be assessed based on the extent to which the pilot clinic implements all components of the intervention appropriately, feedback from clinic staff during implementation of the intervention, and feedback from patients during post-intervention interviews. The investigators anticipate that the intervention will be both feasible and acceptable. Feedback from patients and clinic staff will be used to inform intervention modifications for a larger clinical trial. Effect sizes for the pilot STEPPT intervention (intervention) in comparison to standard care (control) will be assessed by evaluating changes in ethnic disparities (Hispanic vs. Non-Hispanic White) in physician referral to physical therapy and patient adherence to physical therapy referral for the treatment of spine pain before and after implementation of the pilot STEPPT intervention. In comparison to standard care, the investigators expect STEPPT to reduce ethnic disparities in referral and adherence outcomes.

DETAILED DESCRIPTION:
STEPPT is a health system, quality improvement intervention for Hispanic patients with spine pain including the following components: (1) education of providers and staff on disparities in referrals and the benefits of physical therapy for spine pain, (2) modifications to the EHR to automate physical therapy referral and delivery of culturally tailored patient education materials, and (3) enhanced patient health navigation to educate patients and address barriers to attending physical therapy for Hispanic patients with spine pain. This pilot study aims to test the feasibility and acceptability of a prototype intervention developed using patient feedback, focus groups, and collaboration with Family Health Centers of San Diego (FHCSD) administrators and staff. The primary outcome is change in relative rates of referral and adherence to physical therapy between Hispanic and Non-Hispanic White patients with spine pain before and after implementation of the STEPPT intervention within one pilot clinic in the health system. The study will collect data on physical therapy referrals and adherence from electronic health records (EHR) before (3-month usual care control phase) and after (3-month intervention phase) implementing STEPPT. A process evaluation will be conducted through monthly audits and structured observations of clinic workflow. Ongoing interactions with clinic staff will facilitate implementation of the intervention and solicit suggestions for improving feasibility. Post-intervention interviews with a subset of Hispanic patients will assess acceptability of the intervention. Interviews will focus on patient experiences with education materials and enhanced healthcare navigation

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older.
* Patients seeking care within the designated Federally Qualified Health System Adult or Adult Walk-in primary care clinic
* Ethnicity/Race: Participants must identify as either Hispanic or Non-Hispanic White ethnicity/race.
* Consent: Participants must have signed a broad consent for the use of de-identified health information for research.
* Spine Pain: Participants must meet one of the following:

  * New Spine Pain Problem: A new ICD code for neck or back pain added to the problem list during a visit with a primary care physician.
  * Existing Spine Pain Diagnosis: An existing ICD code for neck or back pain on the problem list that is associated with a physician referral for any service during the visit related to the neck or back pain problem.

Exclusion Criteria:

* Non-Musculoskeletal Spine Pain: Participants with spine pain due to a non-musculoskeletal etiology (e.g., infection, cancer, urological disorders, pregnancy) are excluded.
* Urgent Medical Conditions: Patients requiring urgent medical intervention (e.g., fracture, cauda equina syndrome) are excluded.
* Patients with a physical therapy referral external to the healthcare system are excluded from the analysis of physical therapy adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Ethnic Disparity in Rate of Physician Referral to Physical Therapy | 3-month before the intervention and 3 month during intervention period.
  Ethnic disparity (Hispanic vs. Non-Hispanic White) in rate of physician referral of patients with spine pain (low back or neck pain) to physical therapy, as documented in the electronic health record (EHR).
Ethnic Disparity in Rate of Patient Adherence to Physical Therapy Referral | 3-month before the intervention and 3 month during intervention period.
  Ethnic disparity (Hispanic vs. Non-Hispanic White) in rate of attendance of first physical therapy visit after being referred, as documented in the electronic health record (EHR).

SECONDARY OUTCOMES:
Involvement Rating Score | 3-month pilot intervention period.
  Evaluation of clinic staff involvement across various stages of the intervention to assess feasibility and acceptability. Scale values: 0 (min) to 11 (max). Higher values indicate greater involvement in the implementation of STEPPT.
Patient Interviews | Up to 3-months post-intervention
  Qualitative interviews to assess acceptability and potential impact of the STEPPT intervention on Hispanic patients with spine pain.

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Monroe, PT, PhD, Principal Investigator — San Diego State University; Sara Gombatto, PT, PhD, Principal Investigator — San Diego State University
Locations (1):
- Family Health Centers of San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
An IPD sharing plan will be developed for a subsequent stepped wedge clinical trial to assess effectiveness of the final STEPPT intervention. Limited collection of IPD during the developmental phase of this project will not be shared due to time and resource constraints.